CLINICAL TRIAL: NCT05738122
Title: Evaluating the Efficacy of a 60-day Self-guided Emotion Regulation Journal
Brief Title: Evaluating the Efficacy of a 60-day Emotion Regulation Journal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Switch Research (Unknown); Mathematics of Information Technology and Complex Systems (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-0469
Record Dates: First submitted 2023-02-03; First posted 2023-02-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Mental Health; Emotional Regulation
MeSH Terms: conditions — Psychological Well-Being; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Journal Group) (Experimental): Participants in the Intervention group are provided with the 60-day self-guided emotion regulation journals upon enrolment in the study. These participants complete surveys at 2 weeks, 1 month, and 2 months. After the 60-day period, these participants also complete an exit interview and a follow-up survey.
  Interventions: Other: 60-Day self-guided Emotion Regulation Journal
- Control (Waitlist Group) (No Intervention): Participants in the Waitlist group complete a 2-week, 1-month and 2-month survey. After the 60-day period, they receive access to the 60-day self-guided emotion regulation journal for their own use.

INTERVENTIONS:
Other: 60-Day self-guided Emotion Regulation Journal — A 60-day self guided journal with activities designed to be completed daily to improve an individual's emotion regulation abilities and habits
  Arms: Intervention (Journal Group)

SUMMARY:
Participants randomized to the intervention group will receive a physical copy of the 60-day emotion regulation journal during the baseline meeting. Participants will also be introduced the purpose of the journal and its intended usage (i.e., daily journaling). Intervention participants will not be offered guidance or feedback on the journal after these initial instructions, in order to emulate an ad libitum usage. Control group participants will not receive any contact with the researchers outside of the planned questionnaires and to receive their journal at the two-month timepoint.

ELIGIBILITY:
Inclusion Criteria:

* (1) being 18+ years old (2) being fluent in English, (3) currently living in the Greater Victoria area, (4) self-reporting no previously diagnosed mental illness or psychiatric conditions, and (5) scoring a mean of <4.6 on the Cognitive Reappraisal, and mean of >3.14 on the Expressive Suppression subscales of the Emotion Regulation Questionnaire (based on previous mean data)

Exclusion Criteria:

* Scoring a mean of ≥4.6 on the Cognitive Reappraisal or a mean of ≤3.14 on the Expressive Suppression subscales of the Emotion Regulation Questionnaire, currently receiving or seeking therapy for a mental illness, a current or previous diagnosis of mental illness, or self-identifying as neurodivergent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Participant Emotion Regulation | 2 weeks, 1-month, 2-months, 60 day exit interview, 90 days follow up
  Change in participants' emotion regulation abilities and habits assessed using the Emotion Regulation Questionnaire.
Participant Emotion Regulation | 2 weeks, 1-month, 2-months, 60 day exit interview, 90 days follow up
  Change in participants' emotion regulation abilities and habits assessed using the using the Difficulties in Emotional Regulation.

SECONDARY OUTCOMES:
Adherence | 2 weeks, 1-month, 2-months
  Participants' adherence to the 60-days of activities in the journal assessed using three items: "Currently, what is the last day of the journal you have completed?"; "Have you skipped or not completed any days prior to the latest day you have completed?"; and "Approximately how many minutes do you spend completing a day, within the journal?"
Experience using journal | 60 days
  Usability and user experience of intervention group collected during exit interview
Demographics | Baseline
  Age, preferred gender, socio-economic status, ethnicity, educational attainment, and employment status will be collected.
Mental Health | 2 weeks, 1-month, 2-months, and 3-month follow up for intervention group
  Depression and anxiety will be assessed using the Hospital Anxiety and Depression Scale. There is a minimum score of 0 and a maximum score of 21 for each anxiety and depression. Individuals with a score of greater than 8 are considered to have considerable symptoms of anxiety and/or depression.
Subjective Well-Being | 2 weeks, 1-month, 2-months, and 3-month follow up for intervention group
  Subjective well-being will be assessed using the Warwick-Edinburgh Mental Wellbeing Scale. There is a minimum score of 14 and a maximum score of 70. Scores above 51 are above mean population mental well-being while a score below 51 is below mean population mental well-being.
Self-Compassion | 2 weeks, 1-month, 2-months, and 3-month follow up for intervention group
  Self-Compassion will be assessed using the full version of the Self-Compassion Scale. Minimum score is 1 and Maximum score is 5. Scores from 1-2.5 indicate low self-compassion, 2.5-3.5 indicates moderate, and 3.5-5 indicates high self-compassion.
Physical Activity and Sedentary Behaviour | 2 weeks, 1-month, 2-month, and 3-month follow up for intervention group
  Past week hours of sitting, walking, mild, moderate, and vigorous physical activity will be assessed using a modified version of the International Physical Activity Questionnaire. A HIGH score consists of vigorous intensity activity on at least 3 days OR 7 or more days of any combination of walking, moderate intensity or vigorous intensity activities. A MODERATE score consists of 3 or more days of vigorous intensity activity and/or walking of at least 30 minutes per day OR 5 or more days of moderate intensity activity and/or walking of at least 30 minutes per day OR 5 or more days of any combination of walking, moderate intensity or vigorous intensity activities. A LOW score is not achieving the high or moderate physical activity levels.
Screen Time | 2 weeks, 1-month, 2-month, and 3-month follow up for intervention group
  Past week average weekday and weekend occupational and recreational (i.e., leisure) screen time hours will be assessed using four bespoke items (e.g., In the last seven days, on an average weekday, how many hours did you spend using screens for recreational purposes (e.g., watching TV, playing video games)?)
Sleep | 2 weeks, 1-month, 2-month, and 3-month follow up for intervention group
  Past week average hours of sleep will be assessed using an adapted item from the Pittsburgh Sleep Quality Assessment: 20 "During the past week, how many hours of actual sleep did you get at night?". The minimum score is 0 representing 7 or more hours of sleep and the maximum score is 3 representing less than 5 hours of sleep. The higher the score, the worse the sleep duration.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan E Rhodes, PhD, Principal Investigator — University of Victoria
Locations (1):
- Behavioural Medicine Lab - University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No